CLINICAL TRIAL: NCT05402202
Title: Clinical Performance and Accuracy of Healing Abutment With Scan Peg for Single Posterior Implant-supported Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rania Elsayed, Assistant Lecturer, Department of Prosthodontics, Faculty of Dentistry, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IORG0008831
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dental Implants, Single-Tooth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healing abutment with scan peg (Neoss implant system, Harrogate, England) (Experimental): 12 participants will receive Neoss implants by fully-guided implant protocol followed by placement of healing abutment with scan peg
  Interventions: Other: Healing abutment with scan peg (Neoss implant system, Harrogate, England)
- Customized healing abutment (Active Comparator): 12 participants will receive Neoss implants by fully-guided implant protocol followed by placement of customized healing abutment
  Interventions: Other: Customized healing abutment

INTERVENTIONS:
Other: Healing abutment with scan peg (Neoss implant system, Harrogate, England) — 12 participants will receive Neoss implants by fully-guided implant protocol followed by placement of healing abutment with scan peg
  Arms: Healing abutment with scan peg (Neoss implant system, Harrogate, England)
Other: Customized healing abutment — 12 participants will receive Neoss implants by fully-guided implant protocol followed by placement of customized healing abutment fabricated by intraoral scanning by scan body
  Arms: Customized healing abutment

SUMMARY:
The aim of this randomized clinical trial is to evaluate the clinical performance through prosthodontic, periodontal and radiographic evaluation of single screw-retained implant-supported restorations fabricated by intraoral scanning of healing abutment with scan peg in comparison to scan body

DETAILED DESCRIPTION:
Evaluation of the clinical performance through prosthodontic, periodontal and radiographic evaluation of single screw-retained implant-supported restorations fabricated by intraoral scanning of healing abutment with scan peg in comparison to scan body

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are classified as ASA I or II physical status and require mandibular single implants (single missing mandibular posterior teeth) with:

  1. Adequate interarch and mesiodistal space.
  2. Proper bone height and width.
  3. Adequate zone of keratinized tissue (at least 2 mm)

Exclusion Criteria:

1. Any systematic disease as uncontrolled diabetes mellitus or metabolic bone diseases
2. A history of head and neck radiation treatment.
3. Periodontal diseases.
4. Poor oral hygiene (Silness-Löe plaque index score 2 and 3) (32)
5. Parafunctional habits.
6. Malocclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Scanning time (healing abutment-scan peg vs scan body) | Through study completion, an average of 1 year
  The scanning time by intraoral scanner will be recorded in both groups
Quality of proximal contacts of crowns fabricated by intraoral scanning of scan peg vs scan body | Through study completion, an average of 1 year
  The proximal contacts will be evaluated with dental floss
  1. Open: an open contact will be reported if there is no resistance against floss
  2. Ideal: an ideal contact will be reported if there is some resistance to interproximal floss insertion.
  3. Tight: a tight contact will be reported if it prevents the passage of floss through the proximal contact point.
  The percentage of proximal contacts will be calculated for each group at day of crown delivery, 3 months and 6 months later.
Quality of occlusal contacts of crowns fabricated by intraoral scanning of scan peg vs scan body | Through study completion, an average of 1 year
  An evaluation of occlusion will be executed with 2 layers of shim stock of 12µ.
  1. No adjustment: if the shimstock is held when the patient clenches and does not need any adjustment.
  2. Mild adjustment: If the shim stock is held after simple closure, the occlusal contact will be reported as heavy and received mild chairside adjustment.
  3. Major adjustment: If the crown is returned to the manufacturing technician, the adjustment is considered major.
  4. Out of occlusion: If the shim stock passes without resistance after clenching, an open contact will be reported.
  The percentage of occlusal contacts will be calculated for each group at day of crown delivery, 3 months and 6 months later.
Evaluation of occlusion by digital occlusal analyzer | Through study completion, an average of 1 year
  occlusal force of implant-supported restorations will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt